CLINICAL TRIAL: NCT07000019
Title: Combined Aphasia and Robot-Assisted Arm Treatment for Chronic Stroke Survivors
Acronym: CARAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York Medical College (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); New York University (Other)
Responsible Party: Principal Investigator, Tomoko Kitago, MD, Assistant Professor of Neurology, New York Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NYMC-25470; R21DC019955 (NIH)
Record Dates: First submitted 2025-05-23; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Stroke; Aphasia Following Cerebral Infarction; Hemiparesis After Stroke
Keywords: stroke, aphasia, hemiparesis, robotic
MeSH Terms: conditions — Stroke; Aphasia; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined aphasia and robot-assisted arm treatment (Experimental)
  Interventions: Behavioral: CARAT: combined aphasia and robot-assisted arm therapy
- Robot-assisted arm treatment (Active Comparator)
  Interventions: Behavioral: Robot-assisted arm therapy

INTERVENTIONS:
Behavioral: CARAT: combined aphasia and robot-assisted arm therapy — Participants will receive 18 sessions of robot-assisted arm therapy combined with a standardized picture-word verification therapy task with the goal of improving language and arm movements.
  Arms: Combined aphasia and robot-assisted arm treatment
Behavioral: Robot-assisted arm therapy — Participants will receive 18 sessions of robot-assisted arm therapy with the goal of improving arm movements.
  Arms: Robot-assisted arm treatment

SUMMARY:
The goal of this clinical trial is to learn if a program that combines language and arm treatment can improve language and movement problems in people with chronic stroke. The mains questions it aims to answer are:

* To determine the extent to which this combined treatment can improve language.
* To determine the extent to which the combined treatment can improve arm movements.

Researchers will compare the effects of this combined treatment with treatment that targets arm movements alone.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients between 18-90 years of age.
2. Right-handed prior to stroke
3. English-speaking (monolingual)
4. History of single left-hemisphere stroke at least 6 months prior to enrollment
5. Presence of aphasia and naming deficits on Western Aphasia Battery (WAB-R)
6. Comprehension score above 4 on WAB-R
7. Unilateral upper limb paresis (Fugl-Meyer Upper Extremity score <56)
8. Documentation of signed Informed Consent by the study participant.

Exclusion Criteria:

1. Diagnosis or history of speech impairment prior to stroke
2. Severely limited speech output (score below 2 on spontaneous speech portion of WAB-R)
3. Inability to perform screening tasks due to severe language and/or cognitive impairment
4. Condition limiting passive movement in the range of motion required for robotic therapy (e.g. fixed contracture)
5. Any medical or psychiatric condition that may impact participation or compliance with study procedures or activities in the opinion of the investigator

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Philadelphia Naming Test | Baseline to 1 week post-treatment
Fugl-Meyer Upper Extremity Motor Assessment | Baseline to 1 week post-treatment

SECONDARY OUTCOMES:
Western Aphasia Battery-Revised Aphasia Quotient | Baseline to 4 weeks post-treatment
Box and Blocks Test | Baseline to 1 and 4 weeks post-training
Apraxia Battery for Adults | Baseline to 1 and 4 weeks post-training
Stroke and Aphasia Quality of Life Scale-39 | Baseline to 1 and 4 weeks post-training
Apraxia of Speech Rating Scale | Baseline to 1 and 4 weeks post-training

OTHER OUTCOMES:
Arm kinematics | Baseline to 1 and 4 weeks post-training
Arm vs. Non-Arm Naming | Baseline to 1 and 4 weeks post-training

CONTACTS AND LOCATIONS:
Overall Officials: Tomoko Kitago, MD, Principal Investigator — Westchester Medical Center / New York Medical College
Locations (1):
- Westchester Medical Center / New York Medical College, Valhalla, New York, United States

IPD SHARING:
Plan to Share IPD: Yes